CLINICAL TRIAL: NCT01260857
Title: An Open Label, Observational, Post Marketing Surveillance Study To Assess The Safety And Efficacy Of The Spironolactone Plus Hydroflumethiazide (Aldazide) In The Treatment Of Filipino Patients With Stage 1 To 2 Hypertension
Brief Title: Safety And Efficacy Of Spirinolactone Plus Hydroflumethiazide In The Treatment Of Filipino Patients With Hypertension
Status: Withdrawn | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6821003
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Hypertension
Keywords: Spirinolactone; Hydroflumethiazide; Hypertension; Filipinos; Diabetes mellitus; Proteinuria
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Proteinuria | interventions — Hydroflumethiazide

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aldazide — Aldazide 25 mg OD
  Other Names: Spirinolactone + Hydroflumethiazide

SUMMARY:
Aldazide 25 mg OD will be given to Filipino hypertensive patients, and there will be 2 follow-up visits on week 4 and week 8 to monitor for safety and efficacy as primary and secondary outcomes, respectively.

DETAILED DESCRIPTION:
Prospective, non-interventional non-probability sampling

ELIGIBILITY:
Inclusion Criteria:

* Patients >/= 18 years old with Stage 1 or 2 hypertension not controlled by monotherapy or by a combination of anti-hypertensives without any diuretic yet.

Exclusion Criteria:

* Pregnant or lactating women, with hypersensitivity to Aldazide, patients with resistant hypertension not controlled by a combination therapy with a diuretic in their regimen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients ages >/= 18 years old with Stage 1 or 2 hypertension
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Report of Adverse Events occurence (Safety) | 8 weeks

SECONDARY OUTCOMES:
Systolic BP in mmHg | 8 weeks
Diastolic BP in mmHg | 8 weeks
% of patients reaching BP goal of <140/90 mmHg and <130/80 mmHg for DM and proteinuric patients | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6821003&StudyName=Safety%20And%20Efficacy%20Of%20Spirinolactone%20Plus%20Hydroflumethiazide%20In%20The%20Treatment%20Of%20Filipino%20Patients%20With%20Hypertension